CLINICAL TRIAL: NCT02097446
Title: Safety and Efficacy of Antiadhesive Barrier GUARDIX-FL for Women After Laparoscopic Cystectomy : A Prospective, Randomized, Controlled Study
Brief Title: Safety and Efficacy of Antiadhesive Barrier GUARDIX-FL for Women After Laparoscopic Cystectomy
Acronym: GUARDIX-FL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genewel Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Genewel1301
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Genital Diseases, Female
Keywords: cystectomy
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GUARDIX-FL (Experimental): Patients will be treated with 1 or 2 sheet of GUARDIX-FL after ovarian cystectomy(Operative Day).
  Interventions: Device: Guardix-FL
- Interceed (Active Comparator): Patients will be treated with 1 or 2 sheet of interceed after ovarian cystectomy(Operative Day).
  Interventions: Device: Interceed

INTERVENTIONS:
Device: Guardix-FL
  Arms: GUARDIX-FL
Device: Interceed
  Arms: Interceed

SUMMARY:
* Indication: Benign tumors of ovary(mature teratoma, mucinous cystadenoma, serous cystadenoma)
* Intervention: Device ( Test group : Guardix-FL, Control group : Interceed)
* Primary Outcome Measure : Anti-adhesion Rate
* Assessment : Operative Day(Visit 2), Post-Operative Day+7days(Vist 3), Post-Operative Day+4weeks(Visit4), Post-Operative Day+5weeks(Visit 5)

ELIGIBILITY:
Inclusion Criteria:

1. The patients who sign the written informed consent
2. Women aged between 18 and 44
3. The patients who are able to participate in clinical trial during the period of study
4. The patients without abnormal figures at the screening laboratory examination
5. The patients expecting ovarian cystectomy for benign ovarian tumor(mature cystic teratoma, Mucinous cystadenoma, serous cystadenoma)

Exclusion Criteria:

1. The patients who took treatments with medical products which might be barrier to evaluate the effectiveness
2. The patients who took medicine like other anti-adhesion, absorbable hemostat and dose of steroid, immunosuppressants
3. The patients with severe drug allergy
4. The patients with infectious disease on abdominal or pelvic cavity
5. The patients who previously participated in another clinical trials within the past 30 days
6. The patients considered inappropriate for the study
7. The pregnant
8. The patients with severe renal disease
9. The patients with severe systemic diseases

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Anti-Adhesion Rate | Post-Operative Day+4weeks(Second - look)
  Adhesion yes or no

SECONDARY OUTCOMES:
Score | Post-Operative Day+4weeks(Second-look)
  Length of Adhesion x Grade of Adhesion

CONTACTS AND LOCATIONS:
Overall Officials: Joong Sub Choi, Ph.D, Study Director — Hanyang University Seoul Hospital; Seong Hun Kim, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, Seoul, South Korea